CLINICAL TRIAL: NCT06951594
Title: Iowa Cochlear Implant Clinical Research Center Study on Robotic-Assisted Versus Manual Electrode Array Insertion
Brief Title: Robotic-Assisted Versus Manual Electrode Array Insertion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Bruce J Gantz, Chair Emeritus, Department of Otolaryngology--Head and Neck Surgery, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 202210440
Record Dates: First submitted 2025-04-15; First posted 2025-04-30 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: Cochlear Implantation; Robotics
Keywords: cochlear implantation; robotics; hearing preservation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Robot (Experimental): The iotaSOFT™ Insertion System is an FDA approved cochlear implant (CI) electrode array insertion tool. It will be used to assist the surgeon with the cochlear implant insertion.
  Interventions: Device: Robotic
- Manual (No Intervention): Manual cochlear implant surgical procedure without robotic assistance.

INTERVENTIONS:
Device: Robotic — The iotaSOFT™ Insertion System is an FDA approved cochlear implant (CI) electrode array insertion tool. It provides surgeons with consistent insertion speed and force. The system consists of a drive unit connected to a touch screen control console and foot pedal interface. The surgeon secures the base to the skull with two pre-loaded self-drilling bone screws. The drive unit is placed into the base and the adjustable drive head is coupled to a CI electrode. Before insertion begins, the surgeon selects the desired speed of insertion. the surgeon controls the electrode insertion forward and reverse motion via foot pedal while guiding the electrode array into the cochlea with standard CI instrumentation. Upon the completion of electrode array insertion, the drive head and unit are uncoupled from the electrode lead and removed from the patient for disposal.
  Arms: Robot

SUMMARY:
Robotics-assisted electrode insertion overcomes many surgeon-related kinetic limitations such as insertion speed, tremor, drift, and lack of accurate force control. In human cadaveric cochleae, robotics-assisted electrode insertion causes less intracochlear trauma compared to manual insertion. Whether this technical advance results in functional benefits in CI patients remains unknown. To address this critical knowledge gap, the investigators will compare cochlear trauma assessed using CT scans, cochlear and AN function assessed using ECochG and/or the eCAP, and clinical outcomes quantified by postoperative residual acoustic hearing and speech perception scores between participants randomized to either manual or robotics-assisted electrode array insertion.

DETAILED DESCRIPTION:
Electrode insertion force is a critical determinant of the degree/amount of intracochlear trauma caused by CI surgery. It is affected by the speed of electrode array insertion, with higher insertion speeds leading to greater insertion forces. In addition, rapid electrode array insertions with higher forces are associated with translocation of electrode arrays from the scala tympani into the scala media or vestibuli which leads to lower performance and higher rates of loss of residual hearing. Furthermore, variability in insertion force during electrode insertion can cause dramatic increases in intracochlear fluid pressure which appears to be traumatic. The recent FDA-approved iotaSOFT™ insertion system is designed to address these issues by controlling the speed of implant insertion (0.1-1.0 mm/sec) with reduced insertion force and variability. Use of the iotaSOFT™ insertion system significantly reduces the maximum insertion force, variation in insertion force and intracochlear pressure changes over time, which leads to decreased intracochlear trauma compared with manual insertion in cadavers. In addition, this robotics-assisted insertion system can be used with ECochG monitoring systems, which enables response dynamics that can dramatically reduce electrode array stopping distances (1-2 µm of further electrode array advancement) compared to the kinetics of human manual insertion (~1 mm) once a change in intraoperative ECochG response is detected. Theoretically, robotics-assisted electrode array insertion should result in better preserved structural and functional integrity of the peripheral auditory system due to reduced intracochlear trauma. However, this theoretical possibility has not been tested in human CI users.

To address this knowledge gap, the investigators propose to determine the functional benefits of using robotics-assisted electrode insertion in reducing intracochlear trauma. This will be achieved by comparing trauma to the cochlea from electrode insertion based on postoperative CT scans, electrode impedance, the functional status of the cochlea and the AN, as well as preservation of acoustic hearing in participants randomized to have the electrode array inserted manually or with the iotaSOFT™ insertion system. The investigators hypothesize that robotics-assisted electrode insertion will better preserve peripheral structural and functional integrity by reducing intraoperative trauma. The investigators expect that participants with robotics-assisted electrode insertions will show smaller trauma scores based on CT scans, lower electrode impedance, better functional statuses of the AN, higher ENI indices, less hearing loss, and improved speech perception scores than participants with manual electrode insertions.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for a cochlear implant according to CMS guidelines
* Willingness to comply with all study requirements
* Patent cochlea and normal cochlear anatomy, as confirmed by preoperative imaging
* English speaking

Exclusion Criteria:

* Medical or psychological conditions that contraindicate undergoing surgery
* Ossification or any other cochlear anomaly that might prevent complete insertion of the electrode array.
* Unrealistic expectations on the part of the candidate and/or candidate's family, regarding the possible benefits, risks, and limitations that are inherent to the surgical procedure(s) and prosthetic devices.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
scalar translocation | Postoperative standard of care CT (approximately at activation or 2 weeks)
  Postoperative CT scan will be used to assess scalar translocation
Angular Insertion depth | Postoperative standard of care CT (approximately at activation or 2 weeks)
  Angle of the electrode array inside the cochlea, measured relative to the round window membrane.

SECONDARY OUTCOMES:
Impedance | initial activation and at 3 and 6 months post CI
  resistance to the flow of current for each active electrode

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Gantz, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Healthcare, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
Aggregated data will be shared. Individual primary and secondary outcomes are too complex for IPD